CLINICAL TRIAL: NCT02082223
Title: Individualized Preoperative Rehabilitation (iPREHAB) Pilot
Brief Title: Individualized Preoperative Rehabilitation Pilot
Acronym: iPREHAB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Juliane Bingener-Casey, M.D., Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 13-005601
Record Dates: First submitted 2014-03-06; First posted 2014-03-10 (Estimated); Last update posted 2018-02-28 (Actual); Status verified 2018-02

CONDITIONS: Quality of Life; Complex Gastrointestinal Surgery
Keywords: Quality of life; Deficits; Complex gastrointestinal surgery
MeSH Terms: interventions — Immunonutrition Diet; Counseling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Preoperative Rehabilitation (Experimental): Patient & caregiver input regarding 'single biggest concern right now' (modified BEACON buttons) will be elicited. Information gathered by the study team which includes a trained nursing coach and the patient/caregiver will together develop an individualized 'toolbox' of possible interventions to improve preoperative quality of life.
  Candidate interventions include, but not limited to: Participation in SMART program, caregiver participation in Caregivers study protocol MC1295 (IRB 13-002943), nutritional recommendations (deficiencies, immuno-nutrition), low impact resistance training/tai chi, referral to financial or counseling services, establishment of information sources & plans for concerns not frequently covered in clinical practice such as sleeplessness, spiritual assistance.
  Interventions: Behavioral: Interventions to improve preop QOL/resilience deficits

INTERVENTIONS:
Behavioral: Interventions to improve preop QOL/resilience deficits — Identify patients' and patients' care givers quality of life/resilience deficits and supply information and resources prior to undergoing complex GI surgery.
  Other Names: Candidate interventions include, but not limited to:; Participate in SMART (Stress Management And Resiliency Training) program; Caregiver participation in Caregivers study protocol (IRB 13-002943); Nutritional recommendations (deficiencies, immuno-nutrition); Low impact resistance training/tai chi; Referral to financial or counseling services; Establish information sources/plans for concerns not frequently covered in clinical practice such as sleeplessness, spiritual assistance.

SUMMARY:
A pilot to test feasibility of improving patient/caretaker quality of life and resilience.

DETAILED DESCRIPTION:
Our overall goal is to investigate if pre-operative interventions can address patients' and patients' care givers quality of life/resilience deficits and thus improve outcomes. This initial pilot study will test the feasibility of offering patients and their care givers prehabilitation interventions prior to complex gastrointestinal surgery such as pancreatectomy, esophagectomy, proctectomy, or hepatectomy.

ELIGIBILITY:
1. Patients who are being seen for pancreatic, esophageal, rectal or hepatic neoplastic disease, will undergo neo-adjuvant therapy and may require complex GI surgery and their care givers.
2. Are able and willing to participate in all aspects of the study; and
3. Have been provided with, understand the consent.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-03; Primary Completion 2015-06 (Actual); Study Completion 2017-12-25 (Actual)

PRIMARY OUTCOMES:
Feasibility | 3 months post surgical
  Primary outcome is the feasibility of the interventions as measured through the end of study feedback form.

CONTACTS AND LOCATIONS:
Overall Officials: Juliane Bingener-Casey, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States